CLINICAL TRIAL: NCT03047018
Title: Open Trial Investigation of the CHANGE (Changing Health in Autism Through Nutrition, Getting Fit and Expanding Variety) Obesity Program
Brief Title: Open Trial Obesity CHANGE Program ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William Sharp, PhD, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00090911
Record Dates: First submitted 2017-02-07; First posted 2017-02-08 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Autism Spectrum Disorder; Obesity
Keywords: Nutrition
MeSH Terms: conditions — Autism Spectrum Disorder; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHANGE Program (Experimental): Participants with ASD will complete the The Changing Health in Autism through Nutrition, Getting fit and Expanding variety (CHANGE) program.
  Interventions: Behavioral: The Changing Health in Autism through Nutrition, Getting fit and Expanding variety (CHANGE) Program

INTERVENTIONS:
Behavioral: The Changing Health in Autism through Nutrition, Getting fit and Expanding variety (CHANGE) Program — The CHANGE program is a a six-month long intervention consisting of 16 sessions. The first 10 sessions occur weekly while the remaining 6 sessions occur bi-weekly. Sessions last about 1 hour each. Nutrition intervention focuses on decreasing excess calories from liquids and solids and creating a balanced meal plan. Physical activity intervention uses fading strategies to increase participation in exercise. Behavior strategies promote success with meeting goals. Problem-solving techniques address challenges to adherence with implementing the program in the home setting. The standardized protocols include educational handouts, clinic-based activities and assessment procedures, and caregiver-directed homework and data collection.

SUMMARY:
The purpose of this study is to determine if a program can help children with autism who are overweight. Specifically, this study will look to see if changes in a child's eating habits and exercise can help with weight loss. Investigators also want to see how parents feel about the program and if they will complete the entire program.

Twenty children with autism spectrum disorder (ASD) who are also overweight will participate in this study at the Marcus Autism Center. All children who enroll will receive the The Changing Health in Autism through Nutrition, Getting fit and Expanding variety (CHANGE) program. This involves 16 sessions over six months. After the six months, participants will come back every month for three months for a follow up visit. Therefore the study will last a total of nine months.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a program can help children with autism who are overweight. Specifically, this study will look to see if changes in a child's eating habits and exercise can help with weight loss. Investigators also want to see how parents feel about the program and if they will complete the entire program.

This is a 24-week, open trial pilot of 20 children (ages 5 to 12 years old) with ASD and obesity. Subjects will be enrolled in the CHANGE program, a six-month long intervention consisting of 16 sessions. The first 10 sessions occur weekly while the remaining 6 sessions occur bi-weekly. Sessions last about 1 hour each. After 24 weeks, subjects will be asked to return for follow up assessments at 1, 2 and 3 months later.

The primary aims of this project are to 1) determine the feasibility of the intervention, 2) examine preliminary efficacy, and 3) obtain feedback from parents to improve the effectiveness of the intervention and fit for families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ASD using DSM-5 criteria, and clinically significant SCQ score.
* Children with mild to moderate food selectivity, as reflected by a) a diet involving at least 6 food items, b) accepting at least one fruit or vegetable as measured by the Food Preference Inventory (FPI), and c) engaging in low mealtime behavior problems on Brief Autism Mealtime Behavior Inventory (BAMBI) Food Refusal subscale
* Child with a clinic-confirmed body mass index (BMI) percentile in the obese range (i.e., > 95th percentile)
* Parent (primary caregiver) who agrees to participate and attend treatment sessions
* Participating parent able to speak, understand, read, and write in English (assessments, curriculum materials and instructions are in English)

Exclusion Criteria:

* Children with severe feeding problems (e.g., < 5 preferred foods as measured by the FPI) or complex medical issues (e.g., gastrostomy-tube or formula dependent) who require a different treatment approach
* Children on medication associated with weight gain in ASD (e.g., risperidone) that has not yet stabilized (stability criteria defined as 6 months or longer i.e. child has been on medication for less than 6 months).
* Children with serious behavioral problems (i.e., aggression, tantrums, self-injury) or another psychiatric condition that requires a different treatment approach.
* Children with unstable medical conditions or those with a known associated with weight problems will not be included in this study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Willingness to Participate | Baseline through Week 36 Follow Up
  Willingness to participate is measured as <30% refusal of study participation from eligible participants. Willingness to participate will be used to measure overall study feasibility.
Attendance Rate | Baseline through Week 36 Follow Up
  The number of participants who attend all study visits. The attendance rate will be used to measure overall study feasibility. A successful attendance rate will be measured as >70% attendance.
Percent Homework Adherence | Baseline through Week 36 Follow Up
  The percentage of participants who complete all homework assignments. Percent homework adherence will be used to measure overall study feasibility. A successful adherence percentage will be measured as >70%.
Percent Demonstration of Skills | Baseline through Week 36 Follow Up
  The percentage of participants who demonstrate skills learned through the CHANGE program. Percent demonstration of skills will be used to measure overall study feasibility. A successful percentage will be measured as >80%.
Attrition Rate | Baseline through Week 36 Follow Up
  The number of participants who do not complete all study visits. The attrition rate will be used to measure study feasibility. An acceptable attrition rate will be considered <15%.
Percent Satisfaction | Baseline through Week 36 Follow Up
  The percentage of participants who report being satisfied with the intervention. Percent satisfaction will be used to measure overall study feasibility. A successful percentage will be measured as >90%.
Therapist Fidelity to the Treatment Manual | Baseline through Week 36 Follow Up
  The percentage of therapists who adhere to the treatment manual. Therapist fidelity will be used to measure overall study feasibility. A successful percentage rate is >80%.

SECONDARY OUTCOMES:
Difference in Body Mass Index (BMI) Percentile | Baseline through Week 36 Follow Up
  The body mass index is a value derived from the mass and height of an individual. The BMI is defined as the body mass divided by the square of the body height.
Change in Food Preference Inventory (FPI) Score | Baseline through Week 36 Follow Up
  The FPI is a 154-item, parent-reported measure of food selectivity. This measure provides important information about which foods the child eats across food groups. A food selectivity score is calculated by dividing the number of foods rated "never" by the total number of foods listed.
Change in physical activity | Baseline through Week 36 Follow Up
  Physical activity will be measured by parent report and average number of steps by Fitbit data.
Change in Parenting Stress Index- Short Form (PSI-SF) Score | Baseline through Week 36 Follow Up
  The PSI-SF is a 36-item survey commonly used measure parental stress. A higher score indicates more parental stress.

CONTACTS AND LOCATIONS:
Overall Officials: William Sharp, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No